CLINICAL TRIAL: NCT04266717
Title: A Novel Parent Education Program for Early Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Collaborators: Christiana Care Health Services (Other); National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Michele Lobo, Associate Professor, University of Delaware
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PHYT32228419000; 2U54GM104941-06 (NIH)
Record Dates: First submitted 2019-10-08; First posted 2020-02-12 (Actual); Results first posted 2022-10-31 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Preterm Infant; Full-term Infant
Keywords: development; infant; preterm; parent education; play; full-term
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baby Play Parent Education Group (Experimental): Baby Play Intervention involves teaching parents targeted ways they can handle, position, and play with young infants that aim to provide infants enhanced early opportunities to learn to control their bodies and interact with objects. These abilities are associated with future motor, cognitive, and language outcomes. Parents will be asked to perform the intervention activities 20 minutes daily and to log their activity performance weekly.
  Interventions: Behavioral: Baby Play Intervention
- Milestone Education Group (Active Comparator): Parents in the Milestone Education Intervention group will receive information regarding milestones expected based on infants' CA. This information is based on forms from the Centers for Disease Control and Prevention (CDC) and The American Academy of Pediatrics (AAP). This will help parents understand the milestones typically observed at the their child's CA and reflects the education parents receive from healthcare providers. Parents will be asked to provide their infants opportunities to perform these milestone behaviors 20 minutes daily and to log their activity performance weekly.
  Interventions: Behavioral: Milestone Education

INTERVENTIONS:
Behavioral: Baby Play Intervention — Baby Play Intervention involves teaching parents targeted ways they can handle, position, and play with young infants that aim to provide infants enhanced early opportunities to learn to control their bodies and interact with objects. These abilities are associated with future motor, cognitive, and language outcomes. Parents will be asked to perform the intervention activities 20 minutes daily and to log their activity performance weekly.
  Arms: Baby Play Parent Education Group
Behavioral: Milestone Education — Parents in the Milestone Education Intervention group will receive information regarding milestones expected based on infants' CA. This information is based on forms from the Centers for Disease Control and Prevention (CDC) and The American Academy of Pediatrics (AAP). This will help parents understand the milestones typically observed at the their child's CA and reflects the education parents receive from healthcare providers. Parents will be asked to provide their infants opportunities to perform these milestone behaviors 20 minutes daily and to log their activity performance weekly.
  Arms: Milestone Education Group

SUMMARY:
One in ten infants born in the USA is born preterm before 37 weeks of gestation and 50% of those will have motor and cognitive delays requiring intervention at school age. Because existing assessments do not reliably identify motor and cognitive delays early in development, many infants born preterm do not receive early intervention until they are older and their delays are more pronounced. This project aims to address the need for an effective, affordable, novel early intervention model for the first months of life for preterm infants.

DETAILED DESCRIPTION:
One in 10 children in the United States is born preterm and at risk for disabilities that can impair movement and cognition. Research suggests that targeted early intervention can effectively improve ability and function for these children. However, two key obstacles limit the provision of early intervention services in the first half-year of life. First, the existing diagnostic tools are limited in their ability to identify motor and cognitive delays at early ages. Second, in the medical model there is a lack of understanding of developmental science and how experiences in the first months of life can impact the development of future abilities. In effect, there has been lack of knowledge regarding who should receive early intervention services and what activities should be the focus of those services in infancy.

This project aims to address these challenges by testing the fidelity and short-term efficacy of a novel intervention providing education for parents of preterm infants. The intervention will educate parents on ways to handle, position, and play with their infants to provide infants safe opportunities to explore new ways of moving and controlling their bodies and interacting with objects. Intervention provision will be documented and outcomes will be compared for 20 infants randomized to receive one of two types of developmental education. Pre- and post-assessments will compare motor control in prone, reaching ability, daily positioning practices, and parent-child interactions with toys to determine if there are differences in the short-term effects of the intervention. Intervention will occur for two months with parents logging activity daily. Measures related to dosage and how parents perform the intervention activities will be gathered to assess fidelity of the intervention.

Aim 1: To measure aspects related to fidelity for families participating in the study.

Aim 2: To determine if there is a difference in developmental outcomes for children who receive the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Infant meeting the age criteria
* Access to the internet
* Residence within driving distance of the University of Delaware
* Parental ability to read and communicate in English

Exclusion Criteria:

* Genetic diagnosis
* Progressive diagnosis such as spinal muscular atrophy
* Medical or movement restrictions that would interfere with participation in the study activities

Ages: 1 Month to 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2018-01-17 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michele A Lobo, PT, PhD, Principal Investigator — University of Delaware
Locations (1):
- University of Delaware, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: No
This small data set will serve as pilot data for future grant applications.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Baby Play Parent Education Group | Milestone Education Group
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Baby Play Parent Education Group | Milestone Education Group | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: months] | 3.1 (0.9) | 3.8 (1.9) | 3.5 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 5 | 4 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 8 | 9 | 17
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 7 | 7 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Alberta Infant Motor Scale - Change in Total Percentile Score
Description: We will assess infants using the AIMS, a valid and reliable developmental assessment for 0-18-month-olds. It consists of observation of weight bearing, posture, and antigravity movement in supine, prone, sitting, and standing subscales. Infants will receive scores for each subscale (secondary outcomes) that are summer for a total sum score that will be converted to percentile rank (ranging from 0-100). The change in percentile rank from baseline through 1 month will serve as the primary outcome measure for this study to compare the effects of the two interventions with a higher value representing a greater change and the sign representing the direction of change (i.e., positive means developmental performance improved). The AIMS will be used because the PI has shown it to be a sensitive measure of change for FT infants whose parents received handling and positioning education.
Time Frame: at baseline and 1 month later
Measure: Mean (Standard Deviation); unit: change in percentile rank
Arm/Group | Baby Play Parent Education Group | Milestone Education Group
Number analyzed (Participants) | 10 | 10
change in percentile rank | 10 (16.2) | 0 (8.5)
Statistical Analysis 1: Comparison: Baby Play Parent Education Group vs Milestone Education Group; Test type: Superiority; p = 0.016, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Baby Play Parent Education Group | Milestone Education Group
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-09-15): https://cdn.clinicaltrials.gov/large-docs/17/NCT04266717/Prot_SAP_000.pdf
  • Informed Consent Form (2017-11-27): https://cdn.clinicaltrials.gov/large-docs/17/NCT04266717/ICF_001.pdf